CLINICAL TRIAL: NCT04876274
Title: Social Media-Delivered Patient Education in Enhancing Type 2 Diabetics Self-Management and Attitudes During the COVID-19 Pandemic: a Randomized Controlled Trial in Taiwan
Brief Title: Social Media-Delivered Patient Education in Enhancing Type 2 Diabetics Self-Management and Attitudes During the COVID-19 Pandemic
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Medical University (Other)
Collaborators: Taipei Medical University WanFang Hospital (Other)
Responsible Party: Principal Investigator, LEONG CHENG MAN, Master student, School of Pharmacy, Taipei Medical University, Taipei Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: TMU-LOVE
Record Dates: First submitted 2021-05-05; First posted 2021-05-06 (Actual); Results first posted 2021-12-13 (Actual); Last update posted 2022-03-18 (Actual); Status verified 2022-03

CONDITIONS: Type 2 Diabetes
Keywords: Type 2 diabetes; Self-management; Health education; Attitudes towards diabetes; mHealth; Video education
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Health Education

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Patients in the intervention group received Taipei Medical University (TMU) line-oriented video education and care in addition to usual care
  Interventions: Behavioral: TMU-LOVE
- Control group (No Intervention): Patients in the control group received usual care

INTERVENTIONS:
Behavioral: TMU-LOVE — Patients in intervention group could attend diabetes-related health educational video through the TMU-LOVE platform. Researcher would also send 2-3 videos per week with care massage every 2 weeks to the patients.
  Arms: Intervention group

SUMMARY:
The current study was to develop a software "Line@" based health education program, providing video-based health information and communication between diabetes patients and health-care professionals. This study also evaluated its effectiveness on improving glycemic control, attitude towards diabetes, knowledge about diabetes and self-care for type 2 diabetes patients in Taiwan.

The followings were the hypotheses of the study:

1. Compared to the control group, intervention group receiving "Line" based video education has a greater improvement on glycosylated hemoglobin (A1C).
2. Compared to the control group, intervention group receiving "Line" based video education has a greater positive effect on attitude towards diabetes.
3. Compared to the control group, intervention group receiving "Line" based video education has a better understanding on diabetic knowledge.
4. Compared to the control group, intervention group receiving "Line" based video education has a greater positive effect on self-care activity.

DETAILED DESCRIPTION:
The study was conducted in the Endocrinology and Metabolism Clinic in Taipei Medical University Wang-Fang Hospital. Patients were referred from physicians if they met the inclusion criteria and consent to join. Written consent and questionnaires were then provided to the participants after researcher had clearly explained the study purpose.

Based on the seven key points in managing diabetes developed by the association of diabetes care and education specialist (ADCES), including healthy coping, healthy eating, being active, monitoring, taking medication, problem solving and reducing risks, the research team had developed 51 diabetes related health educational videos (available at website of School of Pharmacy, Taipei Medical University http://pharmschool.tmu.edu.tw/activity/index.php?type=20). Each video lasted for about 2-3 minutes. According to the content of the videos, it was categorized into 5 domains, including understanding diabetes, daily care, nutrition care, diabetes drug and diabetes knowledge related quizzes.

Patients in intervention group could attend the video through the line platform. Researcher would also send 2-3 videos per week with care massage every 2 weeks to the patients. The general schedule of video was shown in table x. According to various condition, researcher developed specific video schedule for each patients. For example, patient who was prescribed with A drug, we would only send the video regarding A drug to this patient but not all of the video regarding drugs. Schedule for the part of understanding diabetes, daily care, nutrition care and quizzes was the same among all participants. Due to the quizzes that were put in week 3, 6, 9 and 12, videos related to general knowledge about diabetes would be send to patients first to make sure all the quizzes related content had already taught to patients before the quizzes. Moreover, patients could communicate with the research team and ask questions through the platform, researcher would provide answers verified by pharmacists or physicians in one or two days after.

The sample size of this study was estimated using G-power (version 3.1). Assuming a power of 80% with two-sided alpha level for detecting the difference between the intervention group and the control group, at least 64 patients were needed for each group. Considering 20% dropout rate, the study was designed to have at least 80 patients for each group, 160 patients in total.

Patients were randomized in a 1:1 ratio according to the random allocation sequence generated prior to the study. Patients with odd number were allocated into control group while even numbers were allocated into intervention group. The trial was non-blinded because of its feasibility.

Researcher would not provide any inductive explanation to the patient during filling the questionnaire. If patient had questions about the items, a detailed explanation and health education were provided only after finishing the post-test. The returned questionnaires were collected by the researcher and kept in the Department of Clinical Pharmacy, School of Pharmacy, Taipei Medical University for three years.

All the data were analyzed using SPSS (SPSS Inc. Released 2009. Predictive Analytics Suite Workstation (PASW) Statistics for Windows, Version 18.0. Chicago: SPSS Inc.). A two-tailed p value of 0.05 was considered to be statistically significant in the analysis. For personal characteristics, descriptive analysis was performed. According to the characteristic of data, Chi-square test and t-test was used for detecting the differences between groups. a Wilcoxon signed rank test or paired t-tests was performed for the differences in A1C and the scores between pre and post-test about knowledge, self-care activity and attitude towards diabetes. A Mann-Whitney test or unpaired t-tests was performed for the mean differences between control and intervention group. Logistics regression was performed for the correlation between variables.

Patients who had finished both pre- and post-assessment would be included for analysis, those without post-test would be excluded. Missing values were processed by multiple imputation.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 Diabetes mellitus (T2DM)
* Age 20 or older
* Had at least 1 A1C data in the past 6 months
* Possessed a smart-cellphone
* A1C ≥ 6%

Exclusion Criteria:

* Gestational diabetes
* Cognitive impairment
* No medication treatment but dietary control alone

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 181 (Actual)
Dates: Start 2020-07-14 (Actual); Primary Completion 2020-12-29 (Actual); Study Completion 2020-12-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chen Hsiang-Yin, Pharm.D., Study Director — Professor and Associate Dean, College of Pharmacy, Taipei Medical University
Locations (1):
- School of Pharmacy, Taipei Medical University, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Leong CM, Lee TI, Chien YM, Kuo LN, Kuo YF, Chen HY. Social Media-Delivered Patient Education to Enhance Self-management and Attitudes of Patients with Type 2 Diabetes During the COVID-19 Pandemic: Randomized Controlled Trial. J Med Internet Res. 2022 Mar 23;24(3):e31449. doi: 10.2196/31449. PMID 35319478

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Before assignment, patients were excluded if they did not meet the inclusion criteria or declined to participate, or did not sign the informed consent.
Groups:
- Intervention Group: Patients in the intervention group received the TMU line-oriented video education and care in addition to usual care
  TMU-LOVE: Patients in intervention group could attend diabetes-related health educational video through the TMU-LOVE platform. Researcher would also send 2-3 videos per week with care massage every 2 weeks to the patients.
Period: Overall Study
Arm/Group | Intervention Group | Control Group
Started | 91 | 90
Completed | 82 | 78
Not Completed | 9 | 12
Not completed — Lost to Follow-up | 9 | 12

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention Group | Control Group | Total
Number analyzed (Participants) | 91 | 90 | 181
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.0 (11.4) | 58.1 (11.9) | 58.6 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 33 | 57
  Male | 67 | 57 | 124
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 91 | 90 | 181
Education Level [Count of Participants; unit: Participants]
  Junior high school or below | 14 | 13 | 27
  Senior high school | 26 | 24 | 50
  College or higher | 51 | 53 | 104
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 26.1 (4.2) | 26.7 (5.0) | 26.4 (4.6)
Unemployment [Count of Participants; unit: Participants] | 36 | 40 | 76
Living alone [Count of Participants; unit: Participants] | 3 | 3 | 6
Annual Income (in New Taiwan dollar) [Count of Participants; unit: Participants]
  Unwaged | 28 | 30 | 58
  <500,000 | 18 | 25 | 43
  500,000-1,000,000 | 27 | 21 | 48
  >1,000,000 | 18 | 14 | 32
Medication Type [Count of Participants; unit: Participants]
  Oral medication only | 68 | 72 | 140
  Insulin only | 8 | 1 | 9
  Both | 15 | 17 | 32
Diagnosis Time [Mean (Standard Deviation); unit: years] | 10.4 (9.0) | 10.3 (8.1) | 10.3 (8.5)
HbA1C [Mean (Standard Deviation); unit: %] | 7.0 (0.8) | 6.7 (0.6) | 6.8 (0.7)
Smoking [Count of Participants; unit: Participants] | 10 | 15 | 25
Alcohol Drinking [Count of Participants; unit: Participants] | 36 | 29 | 65
Self Monitoring Blood Glucose [Count of Participants; unit: Participants] | 37 | 42 | 79
Physical Exercise [Count of Participants; unit: Participants] | 70 | 63 | 133

OUTCOME MEASURES:

1. Primary Outcome: HbA1C
Description: Improvement in glycemic control
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: % of HbA1C
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 91 | 90
% of HbA1C | 7.0 (0.9) | 6.7 (0.7)

2. Secondary Outcome: Score of Diabetes Care Profile-Attitudes Toward Diabetes Scales
Description: The Chinese version of Diabetes Care Profile-Attitudes Toward Diabetes Scales (DCP-ATDS) was used for measuring patients' attitude towards diabetes at baseline and 12 weeks. Each item was rated on a five-point Likert scale, the total score was in the range of 23-115, in which higher scores mean patient had better attitudes towards diabetes.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 91 | 90
score on a scale | 3.8 (0.5) | 3.7 (0.5)

3. Secondary Outcome: Score of Summary of Diabetes Self-Care Activities
Description: The Chinese version of Summary of Diabetes Self-Care Activities (SDSCA) was used for measuring patients' self-care activities at baseline and 12 weeks. Each item was rated from 0 to 7. For patients who were prescribed with either oral medication or insulin injection, the total score ranged from 0 to 63. The total score for patients who were taking both oral and insulin medications ranged from 0 to 70. The mean scores were calculated separately according to the total score ranges. A higher scores mean better self-care behavior.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 91 | 90
score on a scale | 4.0 (1.2) | 3.9 (1.5)

4. Secondary Outcome: Score of Simplified True / False Version of Diabetes Knowledge Scale
Description: The Chinese version of Simplified true/false version of revised Diabetes Knowledge Scale (SDKS) was used for measuring patients' knowledge about diabetes at baseline and 12 weeks. A score of "1" was given if the patient responded with the correct answer and "0" was given for incorrect answer or answered with "Don't know". For patients who were prescribed with insulin treatment, the total score ranged from 0 to 24, for those without insulin treatment, the total score ranged from 0 to 22. The mean scores were calculated separately according to the total score ranges. A higher score indicated higher level of knowledge about diabetes.
Time Frame: 12 weeks
Measure: Mean (Standard Error); unit: correctness
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 91 | 90
correctness | 76.7 (11.7) | 73.2 (12.6)

5. Other Pre Specified Outcome: Score of Newest Vital Sign
Description: The Chinese version of Newest Vital Sign (NVS) was used for measuring patients' health literacy level. A score of "1" was given if the patient responded with the correct answer and "0" was given for incorrect answer. The total score ranged from 0 to 6, with higher scores mean better health literacy level.
Time Frame: 12 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Description: All-Cause Mortality, Serious, and Other [Not Including Serious] Adverse Events were not monitored/assessed.
Groups:
- Intervention: Patients in the intervention group received the TMU line-oriented video education and care in addition to usual care
- Control: Patients in the control group received usual care
Arm/Group | Intervention | Control
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
Limitations include the small sample size with a homogenous population in this study, which created population bias and limited the generalizability of the current study. The result in this study could only predict the short-term effect of TMU-LOVE due to a time restriction of 12 weeks, the long-term effect was not feasible.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-02-10): https://cdn.clinicaltrials.gov/large-docs/74/NCT04876274/Prot_SAP_001.pdf